CLINICAL TRIAL: NCT04948905
Title: Assessment of Sense of Identity in Patients With a Diagnosis of Borderline Personality Disorder Through Autobiographical Memory and the Contents of Self-defining Memories, Compared to a Group of Healthy Individuals. A Pilot Study
Brief Title: Assessment of Sense of Identity in Patients Diagnosed With Borderline Personality Disorder. A Pilot Study
Acronym: MASB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2021/AS-01; 2020-A03352-37 (Registry Identifier: N° ID-RCB)
Record Dates: First submitted 2021-06-17; First posted 2021-07-02 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Borderline Personality Disorder
Keywords: Personality Disorder,; Borderline; Psychology; Self-Identity
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed as having Borderline Personality Disorder: These patients have been diagnosed as having Borderline Personality Disorder according to the Diagnostic and Statistical Manual IV classification after taking the Structured Clinical Interview for DSM-IV Axis I Disorders test.
  Interventions: Other: Evaluation using the Self-Defining Memory Questionnaire
- Healthy Controls (Patients not diagnosed as having Borderline Personality Disorder ): These patients have NOT been diagnosed as having Borderline Personality Disorder according to the Diagnostic and Statistical Manual IV classification after taking the Structured Clinical Interview for DSM-IV Axis I Disorders test.
  Interventions: Other: Evaluation using the Self-Defining Memory Questionnaire

INTERVENTIONS:
Other: Evaluation using the Self-Defining Memory Questionnaire — This questionnaire consists of 3 pages. Page 1 gives a clear, concise definition of a memory that defines the self. This enlightens the subject on what is expected and helps him/her consider the phenomenological characteristics of the Self-Defining Memory. Page 2 recalls the 6 essential characteristics of the Self-Defining Memory. Page 3 allows the practical application of what has been understood about the questionnaire. At least 3 memories are asked of the participants. Each memory is rated as follows : On a scale of 0 - 6 for each of the following emotions, participants note how they feel when recalling each memory. Happy, Sad, Angry, Fearful, Surprised, Ashamed,Disgusted,Guilty, Interested, Embarrassed, Contemptful, Proud. 0 = not at all, 3 = Moderately and 6 = Extremely.
  Participants must then use the same scale to indicate the vividness and importance of the memory.
  They must also note the approximate number of years ago the memory took place (to the nearest whole number).

SUMMARY:
One of the key features and long considered a fundamental element of Borderline Personality Disorder is the disruption of identity. Autobiographical memory is closely linked to the development and maintenance of a coherent, stable sense of self. It enables the individual to understand who he or she is. The investigators hypothesize that individuals diagnosed with Borderline Personality Disorder have a less coherent, stable sense of the self than healthy controls. The aim of the study is therefore to compare the sense of identity between a group of patients diagnosed with Borderline Personality Disorder and a group of healthy individuals (without Borderline Personality Disorder ).

This can be measured by evaluating the content of the self-defining memory using the Self-Defining Memory scale.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have given written consent
* Subject affiliated or beneficiary of a health insurance plan.
* Adult subjects between 25 and 55 years of age
* Oral and written mastery of the French language

Inclusion criteria for the borderline group:

* Subject diagnosed as having borderline personality disorder according to the DSM IV classification

Exclusion criteria for the borderline group:

* Patients without diagnosis of borderline personality disorder according to the DSM IV classification after taking the SCID II (Structured Clinical Interview for DSM-III-R Axis II Disorders) test

Exclusion criteria for the control group:

* Subjects considered Borderline after taking the SCID II (Structured Clinical Interview for DSM-III-R Axis II Disorders) test
* Subjects with a score above 8 on the HADS questionnaire corresponding to questionable symptomatology for anxiety and depressive symptoms.

General exclusion Criteria:

* Subjects under court protection, guardianship or curatorship
* Subjects for whom it is impossible to give informed information
* Subjects participating in a Category 1 or 2 RIPH in the 3 months prior to the study
* Subject refusing to give written consent
* Presence of known neurological disease
* Pregnant or breastfeeding women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 30 patients diagnosed as having Bordeline Personality Disorder 30 healthy controls recruited from a poster Campaign within the various departments of Nîmes University Hospital, France.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Sense of Identity in patients diagnosed with Borderline Personality Disorder according to the results of the Self-Defining Memory questionnaire. | Day 7
  The answers to the Self-Defining Memory questionnaire will be analyzed. At least 3 memories are asked of the participants. Each memory is rated as follows : On a scale of 0 - 6 for each of the following emotions, participants note how they feel when recalling each memory. Happy, Sad, Angry, Fearful, Surprised, Ashamed,Disgusted,Guilty, Interested, Embarrassed, Contemptful, Proud. 0 = not at all, 3 = Moderately and 6 = Extremely.
  Participants must then use the same scale to indicate the vividness and importance of the memory.
  They must also note the approximate number of years ago the memory took place (to the nearest whole number).
Sense of Identity in healthy controls according to the results of the Self-Defining Memory questionnaire. | Day 7
  The answers to the Self-Defining Memory questionnaire will be analyzed. At least 3 memories are asked of the participants. Each memory is rated as follows : On a scale of 0 - 6 for each of the following emotions, participants note how they feel when recalling each memory. Happy, Sad, Angry, Fearful, Surprised, Ashamed,Disgusted,Guilty, Interested, Embarrassed, Contemptful, Proud. 0 = not at all, 3 = Moderately and 6 = Extremely.
  Participants must then use the same scale to indicate the vividness and importance of the memory.
  They must also note the approximate number of years ago the memory took place (to the nearest whole number).

SECONDARY OUTCOMES:
Self-coherence of self-defining memories in patients diagnosed with Borderline Personality Disorder | Day 7
  The TALE (Thinking About Life Experiences) self-questionnaire will be used to evaluate this point. This questionnaire contains 15 items, each to be answered with a 5-point Lickert scale (1 = almost never, 5 = very frequently) with the aim of measuring 3 theoretical functions found in the autobiographic memory:
  * The self-continuity function
  * The social bonding function
  * The directing behavior function
Self-coherence of self-defining memories in healthy controls | Day 7
  The TALE (Thinking About Life Experiences) self-questionnaire will be used to evaluate this point. This questionnaire contains 15 items, each to be answered with a 5-point Lickert scale (1 = almost never, 5 = very frequently) with the aim of measuring 3 theoretical functions found in the autobiographic memory:
  * The self-continuity function
  * The social bonding function
  * The directing behavior function
Phenomenological details of self-defining memories in patients diagnosed with Borderline Personality Disorder | Day 7
  The Memory Characteristics Questionnaire (MCQ) will be used to compare the self-defining memories in each group of patients, Borderline vs. Controls. The MCQ is a self-administered questionnaire for the assessment of phenomenological characteristics of autobiographical memory.
  This measurement tool, comprising 15 items and constructed according to a 7-point Likert scale, can distinguish between memories of events, which contain more sensory and contextual details, from memories of contextual details, from memories of imagined events, which contain more elements relating to cognitive operations.
Phenomenological details of self-defining memories in healthy controls | Day 7
  The Memory Characteristics Questionnaire (MCQ) will be used to compare the self-defining memories in each group of patients, Borderline vs. Controls. The MCQ is a self-administered questionnaire for the assessment of phenomenological characteristics of autobiographical memory.
  This measurement tool, comprising 15 items and constructed according to a 7-point Likert scale, can distinguish between memories of events, which contain more sensory and contextual details, from memories of contextual details, from memories of imagined events, which contain more elements relating to cognitive operations.
Traumas undergone in patients diagnosed with Borderline Personality Disorder: Frequency | Day 7
  The Childhood Trauma Questionnaire (CTQ) will be used to evaluate the frequency of traumas undergone by the patient.
  The CTQ is a self-administered questionnaire of childhood and adolescent abuse. The short version, validated in French by David P Bernstein in 2003, includes 28 items and gives a quantitative estimate of the severity of maltreatment experienced. This self-administered questionnaire is based on a 5-point Likert scale and covers five main dimensions of abuse: physical abuse, sexual abuse, emotional abuse, physical neglect and emotional neglect.
Traumas undergone in healthy controls: Frequency | Day 7
  The Childhood Trauma Questionnaire (CTQ) will be used to evaluate the frequency of traumas undergone by healthy controls.
  The CTQ is a self-administered questionnaire of childhood and adolescent abuse. The short version, validated in French (David P Bernstein et al. 2003), includes 28 items and gives a quantitative estimate of the severity of maltreatment experienced. This self-administered questionnaire is based on a 5-point Likert scale and covers five main dimensions of abuse: physical abuse, sexual abuse, emotional abuse, physical neglect and emotional neglect.
Traumas undergone in patients diagnosed with Borderline Personality Disorder: Type | Day 7
  The Childhood Trauma Questionnaire (CTQ) will be used to evaluate the type of traumas undergone by the patient.
  The CTQ is a self-administered questionnaire of childhood and adolescent abuse. The short version, validated in French, includes 28 items and gives a quantitative estimate of the severity of maltreatment experienced. This self-administered questionnaire is based on a 5-point Likert scale and covers five main dimensions of abuse: physical abuse, sexual abuse, emotional abuse, physical neglect and emotional neglect.
Traumas undergone in healthy controls: Type | Day 7
  The Childhood Trauma Questionnaire (CTQ) will be used to evaluate the type of traumas undergone in healthy controls: The CTQ is a self-administered questionnaire of childhood and adolescent abuse. The short version, validated in French by David P Bernstein in 2003, includes 28 items and gives a quantitative estimate of the severity of maltreatment experienced. This self-administered questionnaire is based on a 5-point Likert scale and covers five main dimensions of abuse: physical abuse, sexual abuse, emotional abuse, physical neglect and emotional neglect.

OTHER OUTCOMES:
Age of patients diagnosed with Borderline Personality Disorder | Day 0
  In years
Age of healthy controls | Day 0
  In years
Sex of patients diagnosed with Borderline Personality Disorder | Day 0
  Male/Female
Sex of healthy controls | Day 0
  Male/Female
Level of education of patients diagnosed with Borderline Personality Disorder | Day 0
  The level of education (Primary, Secondary, University, Post-graduate…) will be recorded.
Level of education of healthy controls | Day 0
  The level of education (Primary, Secondary, University, Post-graduate…) will be recorded.
Type of trauma undergone by patients diagnosed with Borderline Personality Disorder | Day 7
  The type of trauma undergone (physical or emotional negligence, physical, sexual or emotional abuse) will be recorded.
Type of trauma undergone by healthy controls | Day 7
  The type of trauma undergone (physical or emotional negligence, physical, sexual or emotional abuse) will be recorded.
Contents of the self-defining memory in patients diagnosed with Borderline Personality Disorder | Day 7
  The contents of the self-defining memory (traumatic memory, neutral memory, pleasant memory) will be recorded.
Contents of the self-defining memory in healthy controls | Day 7
  The contents of the self-defining memory (traumatic memory, neutral memory, pleasant memory) will be recorded.
Other observations in patients diagnosed with Borderline Personality Disorder | Day 7
  Calculated criteria, such as Body Mass Index, based on clinical observations not necessarily found on the case report form may be added to the final database.
Other observations in healthy controls | Day 7
  Calculated criteria, such as Body Mass Index, based on clinical observations not necessarily found on the case report form may be added to the final database.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge LOPEZ-CASTROMAN, Prof., Principal Investigator — Psychiatric Unit, Nîmes University Hospital, France; Stéphane RAFFARD, Prof., Study Director — Montpellier University III, Laboratoire Epsylon, Route de Mende, 34090 Montpellier, France
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France

REFERENCES:
- [Background] Moffitt KH, Singer JA. Continuity in the Life Story: Self-Defining Memories, Affect, and Approach/Avoidance Personal Strivings. Journal of Personality.1994; 62(1), 21-43
- [Background] Singer, J. A., & Moffitt, K. H. An experimental investigation of specificity and generality in memory narratives. Imagination, Cognition and Personality. PsycINFO Database Record (1991-1992)11(3), 233-257.
- [Background] Bluck S, Alea N. Crafting the TALE: construction of a measure to assess the functions of autobiographical remembering. Memory. 2011 Jul;19(5):470-86. doi: 10.1080/09658211.2011.590500. PMID 21864212
- [Background] Johnson MK, Foley MA, Suengas AG, Raye CL. Phenomenal characteristics of memories for perceived and imagined autobiographical events. J Exp Psychol Gen. 1988 Dec;117(4):371-6. PMID 2974863
- [Background] Bernstein, D. P., Fink, L., Handelsman, L., & Foote, J. Childhood Trauma Questionnaire (CTQ) [Database record].(1994) APA PsycTests. https://doi.org/10.1037/t02080-000
- [Background] Spitzer, Robert L, Williams Janet BW, Gibbon Miriam, First Michael B, Structured Clinical Interview for DSM-III-R Axis II Disorders,(SCID-II), Washington, D.C.: American Psychiatric Press, Inc., 1990